CLINICAL TRIAL: NCT04046562
Title: Pain and Weight Treatment: Development and Trial of PAW
Acronym: PAW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Melissa Santos, Principal Investigator, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-079; 1R21DK117221 (NIH)
Record Dates: First submitted 2019-06-07; First posted 2019-08-06 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Adolescent; Pain, Chronic; CBT
MeSH Terms: conditions — Pediatric Obesity; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two arms. One arm is PAW plus standard of care and the second arm is pain education plus standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAW plus standard of care (Active Comparator): Each PAW session will include handouts and worksheets to assist with new strategies as well as homework. Strategies taught within PAW will be integrated with the skills taught in weight management. For example, pain diaries will be kept along with food and exercise logs to examine relationships among pain, eating and activity.
  Interventions: Behavioral: PAW
- Pain education plus standard of care (Placebo Comparator): For those randomized into the information-only group, sessions will be delivered in the same manner. Sessions will cover general pediatric pain management but no behavioral or cognitive skills training will be taught.
  Interventions: Behavioral: Pain Education

INTERVENTIONS:
Behavioral: PAW — Pain and Weight Treatment plus standard of care
  Arms: PAW plus standard of care
Behavioral: Pain Education — Pain Education plus standard of care
  Arms: Pain education plus standard of care

SUMMARY:
Pediatric weight management efficacy is impacted by failure to complete treatment protocols and, for those that do complete treatment, a return to unhealthy behaviors. This project tests whether treating pain, a common comorbid condition to pediatric obesity, will enhance treatment. This study will generate results that can be translated into immediate improvements in care for families seeking treatment for pediatric obesity.

DETAILED DESCRIPTION:
Childhood obesity is a major public health crisis in the United States, affecting 16.9% of youth aged 2-19 and 20.5% of youth aged 12-19. While current family-based interventions are effective in reducing body mass index (BMI) in adolescents; the majority of adolescents regain their excess weight within 2 years. In addition, there is a high rate of drop out from weight management programs, with 27% to 73% of families not completing the full treatment protocol. One possible mechanism influencing pediatric weight management outcomes is chronic pain. Although chronic pain affects 25 to 46% of all youth, among youth with obesity, the prevalence is upwards of 70%. The causal relationship between pain and obesity is not well understood. In some cases, chronic pain may be a precipitant that causes youth to develop obesity by limiting their activities or altering their eating habits. A more common scenario is that obesity places mechanical stresses on the body that can cause pain. With time, pain may become "centralized." Either mechanism may impact youth's participation in a weight management program. However, interventions that address the relationship between chronic pain and obesity in youth are needed, yet no such interventions exist. We expect that co-treating these conditions -obesity and pain- rather than treating just the obesity, will lead to improved pediatric weight management outcomes. The proposed study will take place at the Pediatric Obesity Center at Connecticut Children's Medical Center (CCMC), as an adjunct to our Fit5 program. Fit5 is CCMC's family-based, group weight management treatment program for youth between the ages of 10-18. Consisting of 13 sessions, this multidisciplinary program focuses on behavior changes, nutrition education and physical activity within a cognitive behavioral therapy (CBT) framework. A brief 4 session adjunctive CBT intervention, Pain and Weight treatment (PAW), will be trialed in a group of youth entering weight management treatment and endorsing musculoskeletal pain. This will be done in three phases. First a focus group will be held to review the PAW curriculum which has already been created for this study. In phase two, a small randomized (n = 25 per condition) controlled trial (RCT) will be conducted to pilot PAW. Finally, exit interviews to obtain preliminary feasibility, acceptability and retention data on PAW as compared to an information only control condition will be conducted. There is much work that continues to be needed to improve treatment for youth with obesity. The findings of this study will advance a line of research much needed to better understand outcomes and treatment for adolescents with obesity by shifting from focusing on obesity as an independent condition, and instead, treating it in the context of its comorbid conditions that may be important determinants of engagement, adherence, and outcomes. This proposal will focus on pain and obesity as a model with the intention that this could expand to other comorbidities such as sleep disturbances. The pilot data obtained through this R21 grant proposal will be used to modify the intervention and to seek R01 funding to support a large scale RCT of PAW.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 12 and 18 years of age
* Ability to speak, write and read English
* A parent or guardian who speaks, writes and reads English
* Signed consent and assent from the child and parent
* Enrollment in a weight management program
* Score greater than 3 on the Pain Burden Inventory at screening (in order to recruit adolescents who experience more than just general aches and pains).
* Youth reporting musculoskeletal pain

Exclusion Criteria:

* Parent or guardian unable to participate
* Patients on weight reducing medications
* Severe psychiatric illness (i.e., suicidal or hospitalization within past 6 months)
* Medical conditions such as Type 1 diabetes

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean difference in session attendance between groups | Through the 13 weeks that comprise fit5
  The number of sessions of fit5 attended will be compared between the group attending PAW and those in the information control group.

SECONDARY OUTCOMES:
The feasibility and acceptability of the PAW intervention will be examined Via exit interviews | At the conclusion of the 13 weeks of the program
  At the exit interviews, we will inquire with families whether 4 sessions felt sufficient, whether they would have liked more or less sessions and when they would have liked sessions scheduled.
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Depressed mood: The Center for Epidemiological Studies Depression Scale for Children (CES-DC)
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Eating behaviors (EAH): Three Factor Eating Questionnaire - R18
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Pain symptoms: The Pain Frequency - Severity - Duration Scale
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Pain symptoms: The Adolescent Pediatric Pain Tool
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Self-confidence: Readiness Ruler
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Eating behaviors: Eating Behaviors Questionnaire
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Behavior: The Pediatric Symptom Checklist 17 item (PSC-17)
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Quality of life: Sizing me up
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Quality of life: Sizing them up
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Pain symptoms: The Child Activity Limitations Interview questionnaire
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Pain symptoms: The Child Activity Limitations Interview questionnaire Parent version
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Pain symptoms: Pain Burden Interview
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Sleep: Adolescent Sleep-Wake Scale
The feasibility and acceptability of the PAW intervention will be examined via self-report psychosocial questionnaires. | At the conclusion of the 13 weeks of the program
  Although not powered to be able to detect clinically significant differences pre and post program completion, as part of standard of care families complete a battery of measures prior to and after their completion in the fit5 program. Family scores on these responses will be examined to see if trends show changes in a meaningful and clinically relevant direction.
  Medical: Youth will have their height, weight, BMI and BMI z-score calculated pre and post program completion as well as an assessment of their medical comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Santos, PhD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
NA - we are not planning on sharing the data

REFERENCES:
- See also: Dr. Santos' Obesity Website — https://www.connecticutchildrens.org/specialties-conditions/obesity-weight-management/weight-management-programs